CLINICAL TRIAL: NCT05217550
Title: Veggie Brek: The Feasibility and Acceptability of Offering Vegetables to Children at Breakfast Time in a Nursery Setting: Feasibility Cluster and Randomised Controlled Trial
Brief Title: Testing the Veggie Brek Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loughborough University (Other)
Responsible Party: Principal Investigator, Amanda Daley, Professor of Behavioural Medicine, Loughborough University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Veggie Brek 1: F&A Cluster RCT
Record Dates: First submitted 2021-12-16; First posted 2022-02-01 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Nutrition, Healthy

STUDY DESIGN:
Intervention Model Description: Single-centre interventional cluster randomised controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Veggie Brek) (Experimental): Nursery staff will present vegetables (raw carrot and cucumber batons) to children alongside their main breakfast food for five consecutive days every weekday morning for three weeks.
  Interventions: Behavioral: Veggie Brek
- Control (No Intervention): Children will be served their normal breakfast (with no vegetables) across the three-week intervention period.

INTERVENTIONS:
Behavioral: Veggie Brek — Offering vegetables to children at breakfast alongside their main breakfast food for three consecutive weeks (five days a week) between baseline and follow-up weeks where vegetables are also offered to children at breakfast alongside their main breakfast food for five days a week.
  Arms: Intervention (Veggie Brek)

SUMMARY:
This programme of work aims to investigate the feasibility and acceptability to both children and nursery staff of offering vegetables to children at breakfast time at nursery. Research will be completed to assess the feasibility of undertaking a subsequent cluster randomised controlled trial (RCT) on this question.

DETAILED DESCRIPTION:
Children are not eating a sufficient amount of fruit and vegetables to ensure optimal health and development. Interventions are needed to help increase fruit and vegetable intake from the early years of children's lives, to support the development of lifelong healthy eating habits and the acceptance of vegetables as an important element of a normal diet. Vegetables are often refused by young children due to their often-bitter tastes, and so efforts to increase children's intake of vegetables is a health priority. Vegetables are not commonly offered at breakfast time, which reduces the opportunities each day for vegetables to be part of children's routine diets. Therefore, it is important to understand whether children will be willing to eat - or at least try - vegetables when offered alongside a usual breakfast food (e.g., cereal or toast). Preschool children eat many meals in childcare settings therefore nurseries provide an ideal setting in which to test whether the addition of vegetables at breakfast is feasible and acceptable to both children and nursery staff. This research will recruit nurseries in the East Midlands, UK, to investigate whether children and nursery staff are willing and able to offer (and eat) vegetables at breakfast. The study will adopt a feasibility cluster randomised controlled trial design where nurseries will be randomly allocated to deliver the Veggie Brek intervention or usual breakfast every weekday for three weeks. There will be a baseline period and follow-up period of five days where vegetables will be offered to children at breakfast.

Data will also be collected to understand the nursery staff's views on the study and how easy/difficult the study's procedures were to implement (e.g., were instructions clear and could be followed, were there any barriers to offering vegetables at breakfast). This information will be used to inform the feasibility and acceptability of a later trial.

ELIGIBILITY:
Inclusion Criteria:

* Located in the East Midlands and surrounding areas.

Children:

* Aged 18 months - 4 years.
* Weaned onto solid foods and able to self-feed.
* Eat breakfast at their nursery at least one day a week.

Exclusion Criteria:

* Children with any allergies or intolerances to raw carrot or raw cucumber, or with any conditions which impact feeding or eating in relation to this study (i.e., the offering of raw carrots and cucumber to children in a nursery setting) are not able to take part.

Ages: 18 Months to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 285 (Actual)
Dates: Start 2021-10-18 (Actual); Primary Completion 2022-02-18 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Children's willingness to eat vegetables at breakfast as measured by counts of the vegetables eaten | End of week 5
  The primary outcome is the feasibility and acceptability of the Veggie Brek study intervention which includes an assessment of children's willingness to eat vegetables at breakfast.
Nursery staff's ability to follow the protocol as measured by completion of the data collection sheets | End of week 5
  The primary outcome is the feasibility and acceptability of the Veggie Brek study intervention which includes an assessment of nursery staff's ability to follow the study protocol.
Recruitment rate | End of week 5
  The primary outcome is the feasibility and acceptability of the Veggie Brek study intervention which includes an assessment of the recruitment rate (i.e., parents who provide consent for their child to participate in the study).

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Daley, PhD, Principal Investigator — Loughborough University
Locations (1):
- Loughborough University, Loughborough, Leicestershire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Available upon request once the study findings have been published.
Supporting Information: Study Protocol, ICF
Time Frame: Intention to publish date: 01/12/2023
Access Criteria: Anonymous data will be shared with all who request access via email for novel analyses or re-analysis of the study outcomes. This will be administered by Dr Chris McLeod.

REFERENCES:
- [Derived] McLeod CJ, Haycraft E, Daley AJ. Offering vegetables to children at breakfast time in nursery and kindergarten settings: the Veggie Brek feasibility and acceptability cluster randomised controlled trial. Int J Behav Nutr Phys Act. 2023 Mar 28;20(1):38. doi: 10.1186/s12966-023-01443-z. PMID 36978097